CLINICAL TRIAL: NCT07191834
Title: A Study on the Short - Course Treatment Regimen Containing Pretomanid for Diabetes Mellitus Complicated With Rifampicin - Resistant/Multidrug - Resistant Pulmonary Tuberculosis
Status: Not yet recruiting | Type: Observational
Sponsor: Wuhan Pulmonary Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Wuhan Pulmonary H4
Record Dates: First submitted 2025-08-15; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Rifampicin-resistant/Multidrug-resistant Pulmonary Tuberculosis; Type 2 Diabetes Mellitus (T2DM); Pretomanid
Keywords: pretomanid; T2DM; RR/MDR-TB
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- test group: Thirty patients with diabetes mellitus complicated by rifampicin-resistant/multidrug-resistant pulmonary tuberculosis received a 6-month short-course treatment regimen of bedaquiline, pretomanid, linezolid, and moxifloxacin. From the initiation of treatment to the end of the follow-up period, which lasted a total of 48 weeks, the treatment outcomes and adverse events were observed.
- Control group (Group A): Thirty cases of patients with rifampicin-resistant/multidrug-resistant pulmonary tuberculosis without diabetes received a 6-month short-course treatment regimen of bedaquiline, pretomanid, linezolid, and moxifloxacin. From the initiation of treatment to the end of the follow - up period, which lasted for a total of 48 weeks, the treatment outcomes and adverse events were observed.

SUMMARY:
The treatment of rifampicin-resistant/multidrug-resistant pulmonary tuberculosis (RR-TB) is characterized by a long treatment course, a high incidence of adverse reactions, a low cure rate, and a high recurrence rate. This is related to the large number of drugs in the RR-TB treatment regimen, the high incidence of adverse reactions, and the long treatment course, which lead to poor patient compliance. There is an urgent need for new, effective, safe, and short-course anti-drug-resistant regimens. A 6-month short-course oral regimen containing pretomanid was launched in 2020 and was approved for marketing in China in March 2025. Currently, there have been multi-center studies on the treatment of rifampicin-resistant/multidrug-resistant pulmonary tuberculosis with the pretomanid regimen initiated by investigator-initiated trials (IIT) in China, but there are no studies on special populations. The diabetic population belongs to a special population, has a relatively high incidence rate in China, and is at high risk of tuberculosis. During the treatment process, they may be more likely to experience adverse reactions and poor outcomes than ordinary patients. This study is a prospective cohort clinical study. It is planned to enroll patients aged ≥12 years with RR/MTB-TB complicated by diabetes at our center. Guided by the results of rapid molecular drug susceptibility testing, both groups will be treated with a regimen consisting of bedaquiline, pretomanid, linezolid, and moxifloxacin for 6 months. The experimental group will be diabetic patients, and the control group will be non-diabetic patients. The efficacy and safety of the two groups will be evaluated to provide a basis for the treatment of a new short-course drug-resistant regimen for RR/MDR-TB in special populations in China.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation.
* Aged >12 years, and weighing 30 kilograms or more.
* Patients with pulmonary tuberculosis that is resistant to rifampin (RIF) or to both RIF and isoniazid who initiate an BPaL treatment regimen.
* The diabetes group shall include patients who have been diagnosed with diabetes, either previously or currently.
* Fertile women shall not be pregnant, voluntarily undergo a pregnancy test with a negative result, and be willing to use highly effective contraceptive measures from the time of signing the informed consent until three months after the end of the research treatment.
* Fertile men shall use condoms or other methods to ensure effective contraception for their sexual partners.
* Lactating women shall be willing to stop breastfeeding from the time of signing the informed consent until three months after the end of the research treatment.
* Participants shall voluntarily undergo an HIV test. If the result is positive, they shall voluntarily accept antiretroviral therapy.

Exclusion Criteria:

* Previously received treatment with at least one of bedaquiline (BDQ) or delamanid (DLM) for more than 28 days.
* Currently using prohibited medications specified in the research protocol, and the researcher believes that, from the perspective of patient benefit, the priority of continuing to use the medication is higher than participating in this study.
* Known to have had a hypersensitivity reaction to any of the medications in the protocol.
* Currently participating in any other clinical trials of medications.
* At the time of screening, there is a risk of cardiovascular disease: QTcF interval exceeding 480 milliseconds; a history of arrhythmia considered clinically significant by the researcher within 60 days before enrollment, and the researcher believes that participation in the study may increase the risk; decompensated heart failure; grade 3 hypertension without reaching the control target; abnormal thyroid function; abnormal levels of serum calcium, magnesium, or potassium.
* A history of optic neuropathy or peripheral neuropathy, and the researcher believes that progression/deterioration may occur during the study, or the participant is not suitable for the study.
* At the time of screening, there are the following manifestations of liver diseases: active viral hepatitis; decompensated cirrhosis.
* At the time of screening, there is a history of the following kidney diseases or manifestations related to kidney diseases: a history of unstable or rapidly progressive kidney disease; moderate/severe renal impairment or end - stage renal disease; serum creatinine ≥133 μmol/L in men and ≥124 μmol/L in women.
* Other abnormal laboratory test results: hemoglobin level <8.0 g/dL; platelet count <75,000/mm³; absolute neutrophil count <1000/mm³; aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >3×ULN; total bilirubin >2×ULN, or >1.5×ULN combined with other abnormal liver enzymes; albumin <30 g/L.
* The researcher believes that the study participant is unable to complete the study process, or participation in the study is unsafe for the study participant.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: RR/MDR-TB Patients will be divided into two groups based on the presence or diagnosis of diabetes.
  Experimental group: Patients diagnosed with diabetes. Control group: Patients with diabetes excluded.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
End of treatment outcome | 24 and 48 weeks after treatment initiation
  Number of individuals experiencing each tuberculosis treatment outcome (cure, completion, death, failure, lost-to-follow-up), assessed at the end of treatment by a clinician, based on culture results

SECONDARY OUTCOMES:
Incidence of patients have sputum culture conversion rate of mycobacterium tuberculosis within 48 weeks after treatment completion | 12,24,36 and 48 weeks after treatment initiation
Frequency of any adverse events (AEs) and serious adverse events (SAEs) occurring during the treatment period | From the initiation of treatment to the 48 - week follow - up
  Assessed by a clinician based on symptomatology, subjective screening, and/or laboratory findings.

IPD SHARING:
Plan to Share IPD: No